CLINICAL TRIAL: NCT01288300
Title: Health and Faith (Salud y Fe): Community-Based Diabetes Pilot Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-526-A; 1K23DK087903-01A1 (NIH)
Record Dates: First submitted 2011-01-27; First posted 2011-02-02 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comprehensive diabetes self-management intervention (Active Comparator): Diabetes education, self-empowerment training, exercise, patient navigator
  Interventions: Behavioral: Picture good health/Imaginate una buena salud
- Control (Other): Diabetes self-management lecture
  Interventions: Behavioral: Diabetes lecture

INTERVENTIONS:
Behavioral: Picture good health/Imaginate una buena salud — Diabetes education, self-empowerment training, exercise, patient navigator
  Arms: Comprehensive diabetes self-management intervention
Behavioral: Diabetes lecture — Diabetes self-management lecture
  Arms: Control

SUMMARY:
Main objective: To improve diabetes outcomes among Mexican-Americans with diabetes through church-based, culturally tailored, diabetes self-management interventions linked to the local healthcare system.

Specific Aim: To pilot test a church-based, culturally tailored diabetes self-management intervention to improve diabetes outcomes among low-income Mexican-American with diabetes

H1 A church-based diabetes self-care management curriculum partnered with the local healthcare system will improve glycosylated hemoglobin.

H2 A church-based diabetes self-care management curriculum partnered with the local healthcare system will improve systolic blood pressure and low-density lipids.

H3 A church-based diabetes self-care management curriculum partnered with the local healthcare system will improve diabetes related self-efficacy, self-empowerment and self-care management.

DETAILED DESCRIPTION:
Diabetes is a very prevalent and morbid condition affecting Latinos, especially Mexican-Americans in the United States. South Lawndale, a predominately-Mexican neighborhood of Chicago, has a disproportionately high diabetes related mortality rate in comparison to the rest of Chicago and the U.S. Many church-based interventions have shown promise improving health outcomes among minority populations; but data on church-based interventions for Latino populations is scarce. Mobilizing community resources to develop church-based, diabetes self-management interventions may lead to sustainable, culturally tailored interventions, and improve outcomes in Latinos with diabetes. Considering the growth of the Hispanic population and their disproportionate burden of chronic diseases, developing programming aimed at decreasing the health disparities in this population is crucial. Our study proposes to fill this gap.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* able to speak either English or Spanish
* self-report of diagnosis of diabetes by a doctor

Exclusion Criteria:

* cannot give informed consent (e.g. due to intoxication or dementia)
* do not speak English or Spanish
* younger than 18 years old.
* pregnant women
* undergoing hemodialysis or treatment for cancer
* unable to attend 3- and 6-month follow up appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Changes in glycosylated hemoglobin (Hba1c)from baseline at 3 and 6 months | baseline to 6 months
  We will evaluate changes in HbA1c at baseline, at 3 months and then 6 months. We will analyze change in HbA1c from baseline and compare it to the 3 month and 6 month measures.

SECONDARY OUTCOMES:
Changes in systolic blood pressure at baseline, 3 and 6 months | baseline to 6 months
  We will evaluate changes at baseline, at 3 months and then 6 months. We will analyze change from baseline and compare it to the 3 month and 6 month measures.
Changes in low density lipoprotein from baseline to 3 and 6 month follow up | baseline to 6 months
  We will evaluate changes from baseline, at 3 months and then 6 months. We will analyze change from baseline and compare it to the 3 month and 6 month measures
Changes in diabetes self-care from baseline to 3 and 6 months | baseline to 6 months
  We will evaluate changes from baseline, at 3 months and then 6 months. We will analyze change from baseline and compare it to the 3 month and 6 month measures
Changes in diabetes self-empowerment from baseline to 3 and 6 months | baseline to 6 months
  We will evaluate changes from baseline, at 3 months and then 6 months. We will analyze change from baseline and compare it to the 3 month and 6 month measures

CONTACTS AND LOCATIONS:
Overall Officials: Arshiya A Baig, MD, MPH, Principal Investigator — University of Chicago
Locations (3):
- United States (3):
  - Centro de Salud y Esperanza, Chicago, Illinois
  - Our Lady of Tepeyac Church, Chicago, Illinois
  - St. Agnes of Bohemia Church, Chicago, Illinois

REFERENCES:
- [Derived] Baig AA, Stutz MR, Fernandez Pineros P, Benitez A, Gao Y, Quinn MT, Solomon MC, Sanchez-Johnsen L, Burnet DL, Chin MH; Little Village Community Advisory Board. Using photovoice to promote diabetes self-management in Latino patients. Transl Behav Med. 2019 Nov 25;9(6):1151-1156. doi: 10.1093/tbm/ibz082. PMID 31162592
- [Derived] Baig AA, Benitez A, Locklin CA, Gao Y, Lee SM, Quinn MT, Solomon MC, Sanchez-Johnsen L, Burnet DL, Chin MH; Little Village Community Advisory Board. Picture Good Health: A Church-Based Self-Management Intervention Among Latino Adults with Diabetes. J Gen Intern Med. 2015 Oct;30(10):1481-90. doi: 10.1007/s11606-015-3339-x. Epub 2015 Apr 29. PMID 25920468